CLINICAL TRIAL: NCT03846739
Title: Dose-dependent Effects of Oxytocin on the Amygdala and Reward System Vary Between Women and Men
Brief Title: Dose-dependent Effects of Oxytocin on the Amygdala and Reward System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Chair of the Medical Psychology Division and Deputy Chair of the Department of Psychiatry, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PROXY2
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: amygdala; reward; oxytocin; dose; emotion processing; sex differences

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin & Placebo, 6 IU (Active Comparator): Intranasal administration, 6 IU oxytocin nasal spray or placebo. Imaging starting 45 min after nasal spray administration.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo
- Oxytocin & Placebo, 12 IU (Active Comparator): Intranasal administration,12 IU oxytocin nasal spray or placebo. Imaging starting 45 min after nasal spray administration.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo
- Oxytocin & Placebo, 24 IU (Active Comparator): Intranasal administration, 24 IU oxytocin nasal spray or placebo. Imaging starting 45 min after nasal spray administration.
  Interventions: Drug: Oxytocin nasal spray; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal administration, 6, 12, or 24 international units (IU) oxytocin.
Drug: Placebo — The placebo nasal sprays contain identical ingredients except for the peptide itself.

SUMMARY:
The purpose of this study is to determine whether effects of intranasal oxytocin on amygdala and reward system responses vary as a function of treatment dose in women in comparison to men.

DETAILED DESCRIPTION:
The objective of the present study is to determine whether intranasal oxytocin (IN-OXT) effects on blood oxygenation level-dependent functional magnetic resonance imaging (BOLD fMRI) in the amygdala and striatal regions (putamen, nucleus accumbens, caudate, pallidum) vary as a function of dose. In particular, the investigators plan to compare effects of three different IN-OXT doses (6, 12, and 24 international units, IU) on established neural and behavioural correlates of emotion processing in women. Results will be discussed in comparison to a previous study of OXT kinetics in men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Right-handed
* Non-smoker

Exclusion Criteria:

* Current psychiatric or physical illness
* Hormonal contraception
* Psychoactive medication
* MRI contraindication (e.g. metal in body, claustrophobia)
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Neural substrates of emotion processing, measured via blood-oxygen-level dependent signal in the amygdala | 45 min after nasal spray administration
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal in response to emotional face stimuli. The investigators specifically plan to investigate amygdala responses to emotional faces, because previous studies found sex-specific effects of oxytocin on amygdala activation.
Neural substrates of emotion processing, measured via blood-oxygen-level dependent signal in striatal regions (putamen, nucleus accumbens, caudate, pallidum) | 45 min after nasal spray administration
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal in response to emotional face stimuli. The investigators specifically plan to investigate striatal responses to emotional faces to explore sex-specific effects of OXT on reward-related brain activation.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MD, PhD, Principal Investigator — University of Bonn
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuromodulation of Emotion (NEMO) research group — http://renehurlemann.squarespace.com/welcome/